CLINICAL TRIAL: NCT03101722
Title: Effects of Huperzine a on Presbycusis-related Subjective Tinnitus and Cognitive Impairment
Brief Title: Effects of Huperzine a on Presbycusis(Δ,kHz, DB,MMSE, AD)
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Zhijun Bao (Other)
Responsible Party: Sponsor-Investigator, Zhijun Bao, Huadong hospital, Fudan University, Clinical professor of Otolaryngology, Fudan University
Organization: Fudan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: huadong FudanU
Record Dates: First submitted 2017-03-07; First posted 2017-04-05 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Presbycusis; Tinnitus; Cognitive Impairment
Keywords: presbycusis; tinnitus; cognitive impairment; Huperzine A; age-related hearing impairment
MeSH Terms: conditions — Presbycusis; Tinnitus; Cognitive Dysfunction | interventions — huperzine A; Cholinesterase Inhibitors

STUDY DESIGN:
Intervention Model Description: The studies were divided into 2 groups: Control subgroup and huperzine A group.The study is a single-center, randomized, basic treatment and health education controlled trial, with minimized allocation of patients to one of the two groups.
  For the study of tinnitus intervention, there is a 3 to 12 month follow-up.
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Huperzine A intervention (Experimental): Huperzine A intervention: Huperzine A with a dose 0.1~0.2 mg/time, 2 times/day. BTHE：basic treatment and health education
  Interventions: Drug: BTHE and Huperzine A; Other: BETH
- control (Sham Comparator): Participants in the BTHE group will receive advice regarding lifestyle modification, avoiding alcohol and cigarette consumption.
  Interventions: Drug: BTHE and Huperzine A; Other: BETH

INTERVENTIONS:
Drug: BTHE and Huperzine A — huperzine A intervention
  Other Names: acetylcholinesterase inhibitor
Other: BETH — basic treatment and health education

SUMMARY:
To investigate the effects of huperzine A on tinnitus suppression, hearing and cognitive function protection in patients with presbycusis-related subjective tinnitus and cognitive impairment.

DETAILED DESCRIPTION:
This study is a randomized, controlled trial. 60 eligible participants in total will be recruited. Participants in each group will be evenly and randomly assigned to the huperzine A subgroup and control subgroup using simple randomization method. Participants in the treatment subgroup will receive huperzine A (a dose of 0.2 mg/time, 2 times/day) with basic treatment and health education(BTHE), and those in the control subgroup will receive BTHE only. The primary outcome (auditory function) and secondary outcomes (tinnitus, cognitive symptom and quality of life) will be evaluated at baseline, 3-, 6-, 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

(1) 60 to 85 years old; (2) Mild-to-moderate sensorineural hearing loss (the pure tone averaged across octave frequencies between 0.25 to 4kHz of 26-70 dB HL), with subjective tinnitus, subjective cognitive decline or mild cognitive impairment; (3) Able to tolerate huperzine A treatment; (4) more than 3 months' experience of constant tinnitus; (5) Tinnitus Handicap Inventory score values >10; (6) No participation in any other clinical trial in the past 3 months; (7) Able to accomplish relevant tests and follow-up.

Exclusion Criteria:

(1) Conductive hearing loss; (2) current (3+ months) hearing aid(s) user; (3) Dependence due to poor physical activity; (4) Allergic to huperzine A; (5) History of malignancy within 5 years or other serious medical conditions before screening, including severe bradycardia, hypotension, angina, asthma, ileus, renal insufficiency, neurological diseases (e.g. epilepsy), psychiatric disorder (e.g. schizophrenia, severe depression and anxiety); (6) Acute brain trauma and stroke within 2 weeks; (7) history of general pain disorder and the use of pain relief drugs on a regular basis; (8) Patients who have started treatment or made changes in treatment with drugs known to influence tinnitus within 6 weeks before investigation starts. (9) Individuals simultaneously or previously (within 30 days prior to investigation start) participate in a clinical investigation using experimental drugs or devices. (10) Ongoing serious life event; (11) Vision impairment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-05-15 (Actual); Primary Completion 2030-09-15 (Estimated); Study Completion 2030-09-15 (Estimated)

PRIMARY OUTCOMES:
hearing function protection | 1 years
  All participants (including with tinnitus and without tinnitus) will report in the measure.
  Δ value of averaged hearing threshold = re-test threshold - initial threshold, Δ value of averaged hearing threshold ≤ 0 showed good responders, and > 0 showed poor responders.

SECONDARY OUTCOMES:
global cognitive function protection | 1 years
  All participants (including with tinnitus and without tinnitus) will report in the outcome measure.
  ΔMMSE = re-test MMSE - initial MMSE, ΔMMSE< 0 showed poor responders and hearing threshold ≤ 0 showed good responders; and > 0 showed poor responders ΔMMSE≥ 0 showed good responders
special cognitive domains:orientation to time, orientation to place, registration, attention and calculations,recall, language,repetition and complex commands | 1 years
  MMSE scale in different domains (MMSE SCALE, 0-30)
Tinnitus suppression | 1 years
  150 participants with tinnitus will report in the outcome measure. Method 1: tinnitus functional index (0~100，≤25，relatively mild tinnitus; 25~50,significant problems with tinnitus; ≥50, tinnitus severe enough ）. method 2:no effect on tinnitus was showed "0"; symptomatic alleviation was showed "1";and tinnitus disappear was showed "2"

OTHER OUTCOMES:
adverse events related to treatment of Huperzine A | 1years
  All participants (including with tinnitus and without tinnitus) will be observed gastrointestinal side effects (nausea, vomiting diarrhea)in yes or no, dizziness, fatigue and insomnia in yes or no

CONTACTS AND LOCATIONS:
Overall Officials: zhuowei yu, MD, Study Director — Shanghai Institute of Geriatrics and Gerontology, Shanghai Key Laboratory of Clinical Geriatrics, Huadong Hospital, and Research Center of Aging and Medicine, Shanghai Medical College, Fudan University, Shanghai 200040, China.
Locations (1):
- Huadong Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided